CLINICAL TRIAL: NCT05992415
Title: Know Your Pressures NYC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Lisa Hark, PhD, MBA, Professor of Ophthalmic Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ACYY0034
Record Dates: First submitted 2023-07-28; First posted 2023-08-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma; Hypertension; Glaucoma, Suspect; Elevated Blood Pressure
Keywords: Blood pressure (BP); Intraocular pressure (IOP); Optic nerve imaging; Fundus photography; Blood pressure and glaucoma screening; Optical coherence tomography (OCT); Hypertension (HTN)
MeSH Terms: conditions — Glaucoma; Hypertension; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Know Your Pressures NYC is an innovative, type 2 hybrid effectiveness-implementation 2:1 cluster-randomized clinical trial (RCT) design enrolling individuals living in 14 NYCHA developments, home to 19,098 residents in Upper Manhattan. All participants referred for in-office follow-up exams will be scheduled for an initial appointment, followed by an RCT for those referred. Specific aims are guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) Framework.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Ophthalmology Reading Center outcome assessors and investigators will interpret fundus/optic nerve photographs and OCT imaging and will be masked to participants' demographic and clinical information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Virtual Automated Navigator Intervention with Health Education (Active Comparator): Consented participants referred for follow-up to in-office appointments from the 10 NYCHA developments randomized to the Virtual Automated Navigator Intervention with Health Education Arm will receive text messaging support with all aspects of follow-up appointments at either Columbia University Irving Medical Center or Harlem Hospital, specifically appointment scheduling and education about hypertension and/or glaucoma/suspect over a 1 year period.
  Interventions: Other: Virtual Automated Navigator Intervention with Health Education
- Arm 2: Usual Care (Active Comparator): Consented participants referred for follow-up to in-office appointments from the 4 NYCHA developments randomized to the Usual Care Arm will only be scheduled for their initial appointments at either Columbia University Irving Medical Center or Harlem Hospital. They will not receive enhanced support. Scheduling this initial appointment will allow tracking of adherence. Arm 2 represents a realistic choice available for participants following screening over a 1 year period.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Virtual Automated Navigator Intervention with Health Education — Consented participants referred for follow-up to in-office appointments from the 10 developments randomized to the Virtual Automated Navigator Intervention with Health Education Arm will receive text messaging support via REDCAP with all aspects of follow-up appointments at either Columbia University Irving Medical Center or Harlem Hospital, specifically appointment scheduling and education about hypertension and/or glaucoma/suspect over a 1 year period.
  Arms: Arm 1: Virtual Automated Navigator Intervention with Health Education
Other: Usual Care — Consented participants referred for follow-up to in-office appointments from the 4 developments randomized to the Usual Care Arm will only be scheduled for their initial appointments at either Columbia University Irving Medical Center or Harlem Hospital. They will not receive enhanced support. Scheduling this initial appointment will allow tracking of adherence. Arm 2 represents a realistic choice available for participants following screening over a 1 year period.
  Arms: Arm 2: Usual Care

SUMMARY:
Dr. Lisa A. Hark (PI and Study Chair) and an interdisciplinary team have designed "Know Your Pressures NYC" to conduct blood pressure (BP)/glaucoma screenings in adults age 40+ to identify undiagnosed and/or uncontrolled hypertension and/or glaucoma/suspect. For the purpose of this study, individuals will be identified as glaucoma suspects if they have elevated intraocular pressure (IOP) or have features of glaucoma optic neuropathy, as assessed by optical coherence tomography (OCT) and fundus/optic nerve photographs, as interpreted by the masked Reading Center.

DETAILED DESCRIPTION:
Led by Dr. Lisa A. Hark, with support from an interdisciplinary team with experience in ophthalmology, preventive cardiology, primary care, nursing, biostatistics, implementation science, mixed-methods epidemiology, and informatics, Know Your Pressures NYC is an innovative, type 2 hybrid effectiveness-implementation 2:1 cluster-randomized clinical trial (RCT) design enrolling individuals living in 14 NYCHA developments, home to 19,098 residents in Upper Manhattan. All participants referred for in-office follow-up exams will be scheduled for an initial appointment, followed by an RCT for those referred. Specific aims are guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) Framework.

Aim 1: Conduct combined blood pressure (BP) and glaucoma screenings, and subsequent referrals, among adults age 40+ living in NYC affordable housing developments over 4 years.

Estimation: We will estimate, within a 4% margin of error, the detection rates of undiagnosed and/or uncontrolled HTN and/or glaucoma/suspect by assessing BP, IOP, visual acuity, and optic nerve imaging (OCT and fundus photography).

Aim 2: Evaluate the effectiveness of a Virtual Automated Navigator Intervention with Health Education on appointment adherence in participants referred for follow-up in-office exams after BP/glaucoma screenings compared to Usual Care.

1. The primary Implementation outcome measure for Aim 2 is adherence to in-office appointments for those referred for follow-up.
2. The primary clinical effectiveness outcome measure for Aim 2 is detection of undiagnosed and/or uncontrolled HTN and/or glaucoma/suspect confirmed by in-office appointment(s) and will be measured by rates of newly diagnosed and/or uncontrolled cases of HTN and/or glaucoma/suspect in the office over 1 year.

Hypothesis: Participants referred and randomized to the Virtual Automated Navigator Intervention with Health Education Arm will show higher rates of adherence to in-office appointments over 1 year compared to those receiving Usual Care, who will only receive the initial appointment.

Aim 3: Using RE-AIM, assess Reach, Adoption, Implementation, Maintenance and Sustainability at 1-4 years using a mixed-methods study for those screened and referred.

Hypothesis: Assessing implementation outcomes about Reach (% eligible who are screened); Adoption (% screened who require follow-up); and Maintenance (% returning in 1-year) will inform future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 40 and older.
* Living independently in an affordable housing development.
* Have a cell phone that can receive and send text messages (SMS).

Exclusion Criteria:

* Self-reported terminal illness with life expectancy less than 1 year.
* Inability to provide informed consent due to dementia or other reasons.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7085 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to the Initial In-Office Appointment for those Referred to Ophthalmology and/or Primary Care (Implementation Outcome) | 1 year
  The primary implementation outcome measure for Aim 1 is ADHERENCE TO INITIAL IN-OFFICE APPOINTMENT FOR THOSE REFERRED for follow-up and will be measured by attendance at the initial in-office appointment. The initial in-office appointment will be scheduled by the study team at the conclusion of the BP/glaucoma screening. A comparison will be made between participants living in the 10 developments randomized to the Virtual Automated Intervention Arm compared to 4 developments randomized to Usual Care Arm.
Detection of undiagnosed and/or uncontrolled hypertension and/or glaucoma/suspect for those Referred to follow-up confirmed by in-office eye exam (Clinical Effectiveness Outcome) | 1 year
  The primary clinical effectiveness outcome measure for Aim 2 is detection of undiagnosed and/or uncontrolled HTN and/or glaucoma/suspect confirmed by in-office exams and will calculate the proportion of referred participants who attend and are newly diagnosed and/or treated for uncontrolled HTN and/or glaucoma/suspect in the office over 1 year. Uncontrolled BP is defined as >130/80 mmHg and uncontrolled glaucoma/suspect is defined as IOP >24 including an abnormal optic nerve photograph or OCT image. We will compare the proportion of participants by arm with newly diagnosed and/or uncontrolled HTN and/or glaucoma/suspect in the office over 1 year. Participants who request their own eye doctor will be encouraged to make an appointment as soon as possible. These individuals will be excluded from the Outcome analysis for Aim 2.

SECONDARY OUTCOMES:
Follow-up Adherence to Recommended In-office Exams at 1-3 Years (Secondary Implementation Outcome) | 1-3 years
  A secondary maintenance measure is follow-up adherence to recommended in-office appointments for those who are referred and attend the initial appointment to assess access to care sustainability at 1-4 years. Adherence will be assessed annually on the basis of the expected follow-up schedule defined at the index visit for that year if the participant attends. In the first year, the follow-up recommendation given by the primary care provider and/or the ophthalmologist will be classified into 1 of 4 categories: return within 2 months, return in 3 to 4 months, return in 6 months, or return in 12 months. This follow-up recommendation will be translated into the corresponding expected number of visits per year: 6, 3, 2, or 1.
Return Attendance at Blood Pressure/Glaucoma Screenings at 1-3 Years (Secondary Implementation Outcome) | 1-3 years
  All participants will be invited to return to the BP/eye health screenings at 1, 2, and 3-year follow-up intervals to repeat the BP/glaucoma screening. We hypothesize that participants will return at various intervals (1, 2, and/or 3 times) and we want to understand the demographics and clinical characteristics of these participants as well as the frequency of attendance and why they returned and compare to those who did not elect to participate again. The intervals will be 1,2, and 3 years and we will measure the number and percentage of participants who attend the screenings over 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Hark, Principal Investigator — Columbia University Department of Ophthalmology
Locations (1):
- Columbia University Irving Medical Center - 622 W. 168th St. Floor 18, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No